CLINICAL TRIAL: NCT01669096
Title: Evaluation of the Kinetics of mRNA Expression After Two Doses of GSK Biologicals' Candidate Tuberculosis (Tuberculosis) Vaccine GSK 692342 in Healthy Adults
Brief Title: Study in Healthy Adults to Evaluate Gene Activation After Vaccination With GlaxoSmithKline (GSK) Biologicals' Candidate Tuberculosis (TB) Vaccine GSK 692342
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Aeras (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 116777; 2012-002541-37 (EudraCT Number)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Tuberculosis
Keywords: adults; Tuberculosis vaccine; HIV negative; healthy; mRNA expression
MeSH Terms: conditions — Tuberculosis

ARMS (1):
- GSK 692342 Group (Experimental): Healthy male and female subjects, between and including 18 to 50 years of age, who received 2 doses of GSK 692342 vaccine administered intramuscularly in the deltoid region of the arm, at Days 0 and 30.
  Interventions: Biological: GSK Biologicals' investigational TB vaccine GSK 692342

INTERVENTIONS:
Biological: GSK Biologicals' investigational TB vaccine GSK 692342 — 2 doses administered intramuscularly according to a 0, 1 month schedule (Day 0 and Day 30), in the deltoid region of the arm

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of two doses of the TB vaccine administered according to a 0, 1 month schedule. In, addition, blood samples collected at different time points after vaccination will be analysed to see when exactly genes are activated by the vaccine using an assay called mRNA expression profiling. The different methods for mRNA expression profiling using whole blood samples versus Peripheral Blood Mononuclear cell(s) (PBMCs), will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 50 years of age at the time of obtaining informed consent.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Known BCG vaccination or presence of a BCG scar.
* Seronegative for human immunodeficiency virus-1.
* Female of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of screening and the day of first vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose (for corticosteroids, this will mean prednisone ≥ 20 mg/day or equivalent). Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs starting 2 years before the first dose and planned administration during the study.
* Planned administration/administration of a vaccine/product not foreseen by the study protocol within the period starting 30 days before the first dose of study vaccine and ending at the last study visit.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* History of TB disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* QuantiFERON® TB Gold positive test result.
* History of medically confirmed autoimmune disease.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* History of any reaction of hypersensitivity likely to be exacerbated by any component of the vaccine.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08-21 (Actual); Primary Completion 2012-12-06 (Actual); Study Completion 2013-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Background] van den Berg RA, De Mot L, Leroux-Roels G, Bechtold V, Clement F, Coccia M, Jongert E, Evans TG, Gillard P, van der Most RG. Adjuvant-Associated Peripheral Blood mRNA Profiles and Kinetics Induced by the Adjuvanted Recombinant Protein Candidate Tuberculosis Vaccine M72/AS01 in Bacillus Calmette-Guerin-Vaccinated Adults. Front Immunol. 2018 Mar 26;9:564. doi: 10.3389/fimmu.2018.00564. eCollection 2018. PMID 29632533
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK 692342 Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/African American heritage | 10
  White-Caucasian/European heritage | 9
  Asian-East Asian heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: Antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in femtogram per milliliter (fg/mL), as assessed by cytometric bead array (CBA) assay. The reference seropositivity cut-off value was equal to or above (≥) 7047 fg/mL.
Time Frame: At Day 0 prior to Dose 1
Population: The analysis was performed on the ATP cohort for analysis of immunogenicity, which included all evaluable subjects included in the Total Vaccinated cohort who met all eligibility criteria and for whom post-vaccination blood samples were available for the considered timepoint and assay assessed.
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 18
fg/mL | 6279.7 [4624.2 to 8527.7]

2. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 30 post-Dose 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 18
fg/mL | 7035.1 [5089.0 to 9725.5]

3. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 31 post-Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 17
fg/mL | 64288.5 [33671.9 to 122743.5]

4. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 37 post-Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 18
fg/mL | 32710.5 [23747.1 to 45057.0]

5. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 40 post-Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 18
fg/mL | 8851.2 [5250.8 to 14920.4]

6. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 44 post-Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 18
fg/mL | 6755.1 [4939.5 to 9238.0]

7. Primary Outcome: Concentration of Specific Interferon Gamma (IFN-γ) Antibodies Secreted in Serum Samples
Description: as for outcome 1
Time Frame: At Day 47 post-Dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fg/mL
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 17
fg/mL | 7245.0 [5389.6 to 9739.3]

8. Primary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation CD4+/CD8+ T Cells Expressing at Least Two Different Immune Markers
Description: Among immune markers expressed were interleukin-2 (IL-2) and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ) and/or cluster of differentiation 40-ligand (CD40-L) and/or IL-13 and/or IL-17. The analysis of cytokines expression was performed by flow cytometry using intracellular cytokine staining (ICS) on frozen peripheral blood mononuclear cell (PBMCs).
Time Frame: At Day 0 prior to Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  CD4+CD40-L+IL-2+TNF-α+IFN-γ+IL-17+IL-13 | 97.0 [1.0 to 224.0]
  CD8+CD40-L+IL-2+TNF-α+IFN-γ+IL-17+IL-13 | 95.0 [2.0 to 230.0]

9. Primary Outcome: Frequency of M72 Fusion Protein Specific Cluster of Differentiation CD4+/CD8+ T Cells Expressing at Least Two Different Immune Markers
Description: Among immune markers expressed were interleukin-2 (IL-2) and/or tumour necrosis factor-alpha (TNF-α) and/or interferon-gamma (IFN-γ) and/or cluster of differentiation 40-ligand [CD40-L] and/or IL-13 and/or IL-17. The analysis of cytokines expression was performed by flow cytometry using intracellular cytokine staining (ICS) on frozen peripheral blood mononuclear cell (PBMCs).
Time Frame: At Day 60 post-Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  CD4+CD40-L+IL-2+TNF-α+IFN-γ+IL-17+IL-13 | 5200.0 [485.0 to 15302.0]
  CD8+CD40-L+IL-2+TNF-α+IFN-γ+IL-17+IL-13 | 134.0 [54.0 to 635.5]

10. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers (M1 to M 14)
Description: Expressed immune markers combinations for CD4+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M1=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M2=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M3=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M4=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M5=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M6=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M7=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M8=CD4.CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M9=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M10=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M11=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M12=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M13=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M14=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-).
Time Frame: At Day 0 prior -Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M1 | 1.0 [1.0 to 1.0]
  M2 | 1.0 [1.0 to 26.0]
  M3 | 1.0 [1.0 to 1.0]
  M4 | 96.0 [43.0 to 115.0]
  M5 | 1.0 [1.0 to 1.0]
  M6 | 1.0 [1.0 to 14.0]
  M7 | 1.0 [1.0 to 1.0]
  M8 | 1.0 [1.0 to 14.0]
  M9 | 1.0 [1.0 to 1.0]
  M10 | 1.0 [1.0 to 1.0]
  M11 | 1.0 [1.0 to 1.0]
  M12 | 1.0 [1.0 to 13.0]
  M13 | 1.0 [1.0 to 1.0]
  M14 | 14.0 [1.0 to 17.0]

11. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers (M15 to M28)
Description: Expressed immune markers combinations for CD4+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M15=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M16=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M17=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M18=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M19=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M20=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M21=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M22=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M23=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M24=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M25=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M26=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M27=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M28=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-).
Time Frame: At Day 0 prior-Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M15 | 1.0 [1.0 to 1.0]
  M16 | 15.0 [1.0 to 42.0]
  M17 | 1.0 [1.0 to 1.0]
  M18 | 1.0 [1.0 to 1.0]
  M19 | 1.0 [1.0 to 1.0]
  M20 | 13.0 [1.0 to 14.0]
  M21 | 1.0 [1.0 to 1.0]
  M22 | 1.0 [1.0 to 14.0]
  M23 | 1.0 [1.0 to 1.0]
  M24 | 1.0 [1.0 to 43.0]
  M25 | 1.0 [1.0 to 1.0]
  M26 | 1.0 [1.0 to 1.0]
  M27 | 1.0 [1.0 to 1.0]
  M28 | 1.0 [1.0 to 14.0]

12. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers (M29 to M42)
Description: Expressed immune markers combinations for CD4+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M29=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M30=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M31=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M32=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M33=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M34=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M35=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M36=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M37=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M38=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M39=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M40=CD4.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M41=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M42=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+).
Time Frame: At Day 0 prior - Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M29 | 1.0 [1.0 to 1.0]
  M30 | 1.0 [1.0 to 1.0]
  M31 | 1.0 [1.0 to 1.0]
  M32 | 1.0 [1.0 to 227.0]
  M33 | 1.0 [1.0 to 1.0]
  M34 | 1.0 [1.0 to 1.0]
  M35 | 1.0 [1.0 to 1.0]
  M36 | 1.0 [1.0 to 17.0]
  M37 | 1.0 [1.0 to 1.0]
  M38 | 1.0 [1.0 to 14.0]
  M39 | 1.0 [1.0 to 1.0]
  M40 | 1.0 [1.0 to 14.0]
  M41 | 1.0 [1.0 to 1.0]
  M42 | 1.0 [1.0 to 1.0]

13. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers (M43 to M56)
Description: Expressed immune markers combinations for CD4+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M43=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M44=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M45=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M46=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M47=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M48=CD4.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M49=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M50=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M51=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M52=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M53=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M54=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M55=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M56=CD4.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-).
Time Frame: At Day 0 (prior- Dose 1)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M43 | 1.0 [1.0 to 14.0]
  M44 | 1.0 [1.0 to 1.0]
  M45 | 1.0 [1.0 to 14.0]
  M46 | 1.0 [1.0 to 1.0]
  M47 | 1.0 [1.0 to 1.0]
  M48 | 1.0 [1.0 to 1.0]
  M49 | 1.0 [1.0 to 1.0]
  M50 | 1.0 [1.0 to 13.0]
  M51 | 1.0 [1.0 to 1.0]
  M52 | 1.0 [1.0 to 28.0]
  M53 | 1.0 [1.0 to 1.0]
  M54 | 1.0 [1.0 to 13.0]
  M55 | 1.0 [1.0 to 1.0]
  M56 | 48.0 [1.0 to 90.0]

14. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers (M57 to M63)
Description: Expressed immune markers combinations for CD4+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M57=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M58=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M59=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M60=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M61=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M62=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M63=CD4.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+).
Time Frame: At Day 0 (prior to Dose 1)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M57 | 1.0 [1.0 to 1.0]
  M58 | 1.0 [1.0 to 1.0]
  M59 | 1.0 [1.0 to 1.0]
  M60 | 28.0 [6.0 to 56.0]
  M61 | 1.0 [1.0 to 1.0]
  M62 | 13.0 [1.0 to 16.0]
  M63 | 1.0 [1.0 to 25.0]

15. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M1 to M14)
Description: as for outcome 10
Time Frame: At Day 60 post-Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M1 | 1.0 [1.0 to 1.0]
  M2 | 14.0 [1.0 to 28.5]
  M3 | 21.5 [7.5 to 28.5]
  M4 | 990.0 [517.5 to 1344.5]
  M5 | 1.0 [1.0 to 1.0]
  M6 | 7.5 [1.0 to 24.0]
  M7 | 28.5 [13.5 to 152.0]
  M8 | 1830.5 [1084.5 to 3845.5]
  M9 | 1.0 [1.0 to 1.0]
  M10 | 1.0 [1.0 to 1.0]
  M11 | 1.0 [1.0 to 7.5]
  M12 | 142.5 [86.0 to 228.0]
  M13 | 1.0 [1.0 to 1.5]
  M14 | 1.0 [1.0 to 13.5]

16. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M15 to M28)
Description: Expressed immune markers combinations for CD4+/CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M15=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M16=CD4.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M17=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M18=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M19=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M20=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M21=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M22=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M23=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M24=CD4.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M25=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M26=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M27=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M28=CD4.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-).
Time Frame: At Day 60 post - Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M15 | 7.0 [1.0 to 55.5]
  M16 | 1202.5 [561.5 to 1827.5]
  M17 | 1.0 [1.0 to 1.0]
  M18 | 1.0 [1.0 to 1.0]
  M19 | 1.0 [1.0 to 15.5]
  M20 | 300.0 [94.5 to 529.5]
  M21 | 1.0 [1.0 to 1.0]
  M22 | 18.5 [13.5 to 28.0]
  M23 | 1.0 [1.0 to 28.0]
  M24 | 666.5 [230.5 to 1220.5]
  M25 | 1.0 [1.0 to 1.0]
  M26 | 1.0 [1.0 to 1.0]
  M27 | 1.0 [1.0 to 1.0]
  M28 | 87.0 [40.5 to 179.5]

17. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M29 to M42)
Description: as for outcome 12
Time Frame: At Day 60 post Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M29 | 1.0 [1.0 to 1.0]
  M30 | 1.0 [1.0 to 14.0]
  M31 | 1.0 [1.0 to 22.5]
  M32 | 1198.5 [80.5 to 2845.5]
  M33 | 1.0 [1.0 to 1.0]
  M34 | 1.0 [1.0 to 1.0]
  M35 | 1.0 [1.0 to 1.0]
  M36 | 28.0 [1.0 to 78.0]
  M37 | 1.0 [1.0 to 1.0]
  M38 | 1.0 [1.0 to 7.5]
  M39 | 1.0 [1.0 to 1.0]
  M40 | 69.0 [20.0 to 225.5]
  M41 | 1.0 [1.0 to 1.0]
  M42 | 1.0 [1.0 to 1.0]

18. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers,Post Dose 2 (M43 to M56)
Description: as for outcome 13
Time Frame: At Day 60 (post-Dose 2)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M43 | 1.0 [1.0 to 14.0]
  M44 | 1.0 [1.0 to 1.0]
  M45 | 13.5 [1.0 to 18.0]
  M46 | 1.0 [1.0 to 7.5]
  M47 | 66.0 [1.0 to 121.0]
  M48 | 1.0 [1.0 to 1.0]
  M49 | 1.0 [1.0 to 1.0]
  M50 | 1.0 [1.0 to 1.0]
  M51 | 1.0 [1.0 to 1.0]
  M52 | 55.5 [29.0 to 184.0]
  M53 | 1.0 [1.0 to 1.0]
  M54 | 28.0 [7.0 to 36.0]
  M55 | 1.0 [1.0 to 1.0]
  M56 | 163.0 [75.5 to 383.0]

19. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD4+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M57 to M63)
Description: as for outcome 14
Time Frame: At Day 60 post- Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M57 | 1.0 [1.0 to 1.0]
  M58 | 1.0 [1.0 to 13.5]
  M59 | 1.0 [1.0 to 7.5]
  M60 | 15.0 [1.0 to 145.5]
  M61 | 1.0 [1.0 to 1.0]
  M62 | 20.5 [1.0 to 34.0]
  M63 | 1.0 [1.0 to 50.0]

20. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers (M1 to M14)
Description: Expressed immune markers combinations for CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M1=CD8.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M2=CD8.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M3=CD8.CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M4=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M5=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M6=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M7=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M8=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M9=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M10=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M11=CD8.CD40L(+)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M12=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M13=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M14=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+).
Time Frame: At Day 0 prior-Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M1 | 1.0 [1.0 to 1.0]
  M2 | 1.0 [1.0 to 1.0]
  M3 | 1.0 [1.0 to 23.0]
  M4 | 1.0 [1.0 to 1.0]
  M5 | 1.0 [1.0 to 1.0]
  M6 | 1.0 [1.0 to 1.0]
  M7 | 1.0 [1.0 to 1.0]
  M8 | 1.0 [1.0 to 1.0]
  M9 | 1.0 [1.0 to 1.0]
  M10 | 1.0 [1.0 to 1.0]
  M11 | 1.0 [1.0 to 1.0]
  M12 | 1.0 [1.0 to 1.0]
  M13 | 1.0 [1.0 to 1.0]
  M14 | 1.0 [1.0 to 1.0]

21. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers (M15 to M28)
Description: Expressed immune markers combinations for CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M15=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M16=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M17=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M18=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M19=CD8.CD40L(+)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M20=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M21=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M22=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M23=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M24=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M25=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M26=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M27=CD8.CD40L(-)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M28=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+).
Time Frame: At Day 0 prior -Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M15 | 1.0 [1.0 to 1.0]
  M16 | 1.0 [1.0 to 1.0]
  M17 | 1.0 [1.0 to 1.0]
  M18 | 1.0 [1.0 to 1.0]
  M19 | 6.0 [1.0 to 128.0]
  M20 | 1.0 [1.0 to 1.0]
  M21 | 1.0 [1.0 to 1.0]
  M22 | 1.0 [1.0 to 1.0]
  M23 | 1.0 [1.0 to 1.0]
  M24 | 1.0 [1.0 to 1.0]
  M25 | 1.0 [1.0 to 1.0]
  M26 | 1.0 [1.0 to 1.0]
  M27 | 1.0 [1.0 to 1.0]
  M28 | 1.0 [1.0 to 1.0]

22. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers (M29 to M42)
Description: Expressed immune markers combinations for CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M29=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M30=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M31=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M32=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M33=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M34=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M35=CD8.CD40L(-)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(-); M36=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M37=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M38=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M39=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M40=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M41=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-); M42=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+).
Time Frame: At Day 0 prior- Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M29 | 1.0 [1.0 to 1.0]
  M30 | 1.0 [1.0 to 1.0]
  M31 | 1.0 [1.0 to 1.0]
  M32 | 1.0 [1.0 to 1.0]
  M33 | 1.0 [1.0 to 1.0]
  M34 | 1.0 [1.0 to 1.0]
  M35 | 1.0 [1.0 to 62.0]
  M36 | 1.0 [1.0 to 1.0]
  M37 | 1.0 [1.0 to 1.0]
  M38 | 1.0 [1.0 to 1.0]
  M39 | 32.0 [3.0 to 160.0]
  M40 | 1.0 [1.0 to 1.0]
  M41 | 1.0 [1.0 to 1.0]
  M42 | 1.0 [1.0 to 1.0]

23. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers (M43 to M56)
Description: Expressed immune markers combinations for CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M43=CD8.CD40L(-)+IL-2(-)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M44=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M45=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M46=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M47=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M48=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+); M49=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(-); M50=CD8.CD40L(-)+IL-2(-)+TNF-α(-)+IFN-γ(-)+IL-17(-)+IL-13(+); M51=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(+); M52=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(+)+IL-13(-); M53=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(+); M54=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(+)+IL-17(-)+IL-13(-); M55=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(+); M56=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(+)+IL-13(-).
Time Frame: At Day 0 prior to Dose 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M43 | 38.0 [4.0 to 69.0]
  M44 | 1.0 [1.0 to 1.0]
  M45 | 1.0 [1.0 to 1.0]
  M46 | 1.0 [1.0 to 1.0]
  M47 | 66.0 [1.0 to 333.0]
  M48 | 1.0 [1.0 to 1.0]
  M49 | 1.0 [1.0 to 31.0]
  M50 | 1.0 [1.0 to 101.0]
  M51 | 1.0 [1.0 to 1.0]
  M52 | 1.0 [1.0 to 1.0]
  M53 | 1.0 [1.0 to 1.0]
  M54 | 1.0 [1.0 to 1.0]
  M55 | 1.0 [1.0 to 1.0]
  M56 | 1.0 [1.0 to 1.0]

24. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers (M57 to M63)
Description: Expressed immune markers combinations for CD8+ T cells included CD40-L, IL-2, TNF-α, IFN-γ, IL-17 and IL-13, as follows: M57=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(+); M58=CD8_CD40L(+)+IL-2(+)+TNF-α(+)+IFN-γ(-)+IL-17(-)+IL-13(-); M59=CD8_CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(+); M60=CD8_CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(+)+IL-13(-); M61=CD8_CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(+); M62=CD8_CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(+)+IL-17(-)+IL-13(-); M63=CD8_CD40L(+)+IL-2(+)+TNF-α(-)+IFN-γ(-)+IL-17(+)+IL-13(+).
Time Frame: At Day 0 (prior to Dose 1)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 13
T cells/million cells
  M57 | 1.0 [1.0 to 1.0]
  M58 | 1.0 [1.0 to 1.0]
  M59 | 1.0 [1.0 to 1.0]
  M60 | 1.0 [1.0 to 1.0]
  M61 | 1.0 [1.0 to 1.0]
  M62 | 1.0 [1.0 to 1.0]
  M63 | 1.0 [1.0 to 1.0]

25. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M1 to M14)
Description: as for outcome 20
Time Frame: At Day 60 post-Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M1 | 1.0 [1.0 to 1.0]
  M2 | 1.0 [1.0 to 1.0]
  M3 | 1.0 [1.0 to 42.0]
  M4 | 1.0 [1.0 to 1.0]
  M5 | 1.0 [1.0 to 1.0]
  M6 | 1.0 [1.0 to 1.0]
  M7 | 1.0 [1.0 to 10.0]
  M8 | 1.0 [1.0 to 1.0]
  M9 | 1.0 [1.0 to 1.0]
  M10 | 1.0 [1.0 to 1.0]
  M11 | 1.0 [1.0 to 1.0]
  M12 | 1.0 [1.0 to 1.0]
  M13 | 1.0 [1.0 to 1.0]
  M14 | 1.0 [1.0 to 1.0]

26. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M15 to M28)
Description: as for outcome 21
Time Frame: At Day 60 post -Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M15 | 1.0 [1.0 to 1.0]
  M16 | 1.0 [1.0 to 1.0]
  M17 | 1.0 [1.0 to 1.0]
  M18 | 1.0 [1.0 to 1.0]
  M19 | 1.0 [1.0 to 43.5]
  M20 | 1.0 [1.0 to 1.0]
  M21 | 1.0 [1.0 to 1.0]
  M22 | 1.0 [1.0 to 1.0]
  M23 | 1.0 [1.0 to 22.5]
  M24 | 1.0 [1.0 to 1.0]
  M25 | 1.0 [1.0 to 1.0]
  M26 | 1.0 [1.0 to 1.0]
  M27 | 1.0 [1.0 to 1.0]
  M28 | 1.0 [1.0 to 1.0]

27. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M29 to M42)
Description: as for outcome 22
Time Frame: At Day 60 post- Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M29 | 1.0 [1.0 to 1.0]
  M30 | 1.0 [1.0 to 1.0]
  M31 | 1.0 [1.0 to 61.5]
  M32 | 1.0 [1.0 to 1.0]
  M33 | 1.0 [1.0 to 1.0]
  M34 | 1.0 [1.0 to 1.0]
  M35 | 14.5 [1.0 to 110.5]
  M36 | 1.0 [1.0 to 1.0]
  M37 | 1.0 [1.0 to 1.0]
  M38 | 1.0 [1.0 to 1.0]
  M39 | 40.5 [1.0 to 339.5]
  M40 | 1.0 [1.0 to 1.0]
  M41 | 1.0 [1.0 to 1.0]
  M42 | 1.0 [1.0 to 1.0]

28. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M43 to M56)
Description: as for outcome 23
Time Frame: At Day 60 post-Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M43 | 10.0 [1.0 to 189.5]
  M44 | 1.0 [1.0 to 1.0]
  M45 | 1.0 [1.0 to 1.0]
  M46 | 1.0 [1.0 to 1.0]
  M47 | 109.0 [1.0 to 1432.5]
  M48 | 1.0 [1.0 to 1.0]
  M49 | 1.0 [1.0 to 13.0]
  M50 | 13.5 [1.0 to 64.5]
  M51 | 1.0 [1.0 to 1.0]
  M52 | 1.0 [1.0 to 1.0]
  M53 | 1.0 [1.0 to 1.0]
  M54 | 45.0 [1.0 to 57.5]
  M55 | 1.0 [1.0 to 1.0]
  M56 | 1.0 [1.0 to 1.0]

29. Primary Outcome: Frequency of M72 Specific Cluster of Differentiation CD8+ T Cells Expressing Any Combination of Immune Markers, Post Dose 2 (M57 to M63)
Description: as for outcome 24
Time Frame: At Day 60 post Dose 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 12
T cells/million cells
  M57 | 1.0 [1.0 to 1.0]
  M58 | 1.0 [1.0 to 1.0]
  M59 | 1.0 [1.0 to 1.0]
  M60 | 1.0 [1.0 to 1.0]
  M61 | 1.0 [1.0 to 1.0]
  M62 | 1.0 [1.0 to 1.0]
  M63 | 1.0 [1.0 to 1.0]

30. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Month 7)
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Participants | 1

31. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Participants
  Any Pain, Dose 1 | 18
  Grade 3 Pain, Dose 1 | 3
  Any Redness, Dose 1 | 4
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 4
  Grade 3 Swelling, Dose 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 17
  Any Pain, Dose 2 | 15
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 17
  Grade 3 Pain, Dose 2 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 17
  Any Redness, Dose 2 | 4
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 17
  Grade 3 Redness, Dose 2 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 17
  Any Swelling, Dose 2 | 3
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 17
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Across doses | 18
  Grade 3 Pain, Across doses | 3
  Any Redness, Across doses | 4
  Grade 3 Redness, Across doses | 1
  Any Swelling, Across doses | 5
  Grade 3 Swelling, Across doses | 0

32. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were Fatigue, Gastrointestinal symptoms, Headache, Malaise, Myalgia and Fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = incidence of any particular symptom regardless of intensity grade. Grade 3 = incidence of a particular symptom that prevented normal, everyday activity. Grade 3 fever = axillary temperature above (>) 39.5 °C. Related = general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Participants
  Any Fatigue, Dose 1 | 8
  Related Fatigue, Dose 1 | 8
  Grade 3 Fatigue, Dose 1 | 0
  Any Gastrointestinal symptoms, Dose 1 | 3
  Related Gastrointestinal symptoms, Dose 1 | 3
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0
  Any Headache, Dose 1 | 6
  Related Headache, Dose 1 | 6
  Grade 3 Headache, Dose 1 | 0
  Any Malaise, Dose 1 | 7
  Related Malaise, Dose 1 | 7
  Grade 3 Malaise, Dose 1 | 0
  Any Myalgia, Dose 1 | 3
  Related Myalgia, Dose 1 | 3
  Grade 3 Myalgia, Dose 1 | 0
  Any Fever, Dose 1 | 2
  Related Fever, Dose 1 | 2
  Grade 3 Fever, Dose 1 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 17
  Any Fatigue, Dose 2 | 11
  Related Fatigue, Dose 2: number analyzed (Participants) | 17
  Related Fatigue, Dose 2 | 11
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 17
  Grade 3 Fatigue, Dose 2 | 2
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17
  Any Gastrointestinal symptoms, Dose 2 | 4
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17
  Related Gastrointestinal symptoms, Dose 2 | 4
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 17
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 17
  Any Headache, Dose 2 | 11
  Related Headache, Dose 2: number analyzed (Participants) | 17
  Related Headache, Dose 2 | 10
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 17
  Grade 3 Headache, Dose 2 | 2
  Any Malaise, Dose 2: number analyzed (Participants) | 17
  Any Malaise, Dose 2 | 9
  Related Malaise, Dose 2: number analyzed (Participants) | 17
  Related Malaise, Dose 2 | 9
  Grade 3 Malaise, Dose 2: number analyzed (Participants) | 17
  Grade 3 Malaise, Dose 2 | 2
  Any Myalgia, Dose 2: number analyzed (Participants) | 17
  Any Myalgia, Dose 2 | 8
  Related Myalgia, Dose 2: number analyzed (Participants) | 17
  Related Myalgia, Dose 2 | 7
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 17
  Grade 3 Myalgia, Dose 2 | 2
  Any Fever, Dose 2: number analyzed (Participants) | 17
  Any Fever, Dose 2 | 7
  Related Fever, Dose 2: number analyzed (Participants) | 17
  Related Fever, Dose 2 | 5
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 17
  Grade 3 Fever, Dose 2 | 0
  Any Fatigue, Across doses | 14
  Related Fatigue, Across doses | 14
  Grade 3 Fatigue, Across doses | 2
  Any Gastrointestinal symptoms, Across doses | 6
  Related Gastrointestinal symptoms, Across doses | 6
  Grade 3 Gastrointestinal symptoms, Across doses | 0
  Any Headache, Across doses | 13
  Related Headache, Across doses | 13
  Grade 3 Headache, Across doses | 2
  Any Malaise, Across doses | 11
  Related Malaise, Across doses | 11
  Grade 3 Malaise, Across doses | 2
  Any Myalgia, Across doses | 10
  Related Myalgia, Across doses | 9
  Grade 3 Myalgia, Across doses | 2
  Any Fever, Across doses | 8
  Related Fever, Across doses | 6
  Grade 3 Fever, Across doses | 0

33. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related AE = an AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Participants | 12

34. Primary Outcome: Number of Subjects With Potential Immune-Mediated Disease(s) (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (From Day 0 to Month 7)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | GSK 692342 Group
Number analyzed (Participants) | 20
Participants | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period following each dose and across doses; unsolicited AEs: During the 30-day (Days 0-29) post-vaccination period; pIMDs: during the entire study period (From Day 0 to Month 7).
Arm/Group | GSK 692342 Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 692342 Group (N=20)
Alcohol abuse (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK 692342 Group (N=20)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (8)
Fatigue (General disorders) | 14 (19)
Feeling hot (General disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 6 (7)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 13 (19)
Injection site warmth (General disorders) | 1 (1)
Malaise (General disorders) | 12 (17)
Migraine (Nervous system disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12)
Pain (General disorders) | 18 (33)
Pertussis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 8 (9)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Swelling (General disorders) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.